CLINICAL TRIAL: NCT05987722
Title: Effectiveness of Enoxolone on Oral Conditions of Patients With Periodontal Surgery
Acronym: Enoxolone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20200136
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-04

CONDITIONS: Periodontal Surgery
Keywords: Enoxolone; Wound healing; Plaque index.
MeSH Terms: interventions — Glycyrrhetinic Acid; Sensodyne

STUDY DESIGN:
Intervention Model Description: Each patient underwent routine periodontal surgery procedures: (1) On the first day of surgery, the researchers confirmed the correctness of the patient's oral hygiene instructions before surgery; (2) All periodontal surgery was performed by the same dentist. After periodontal surgery was sutured, antibiotics (Amoxicillin 500 mg, every 8 h, for 7 days) and painkillers (Acetaminophen 250 mg, every 6 h as long as it is painful) were provided. The experimental group (N=15) returned home after the operation and used BGA toothpaste (Enoxolone) three times a day for oral cleaning for 12 weeks. The control group (N=12) used BGA-free toothpaste (Sensodyne) for oral cleaning, and the rest of the research time, measurement time and measurement results were the same as those of the experimental group.
Masking Description: The experimental group and the control group were randomly assigned by lottery drawing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxolone (Experimental): The experimental group (N=15) returned home after the operation and used BGA toothpaste (Enoxolone) three times a day for oral cleaning for 12 weeks.
  Interventions: Other: Enoxolone
- Sensodyne (Active Comparator): The control group (N=12) used BGA-free toothpaste (Sensodyne) for oral cleaning for 12 weeks.
  Interventions: Other: Sensodyne

INTERVENTIONS:
Other: Enoxolone — The experimental group returned home after the operation and used glycyrrhetinic acid toothpaste three times a day for oral cleaning.After the operation, toothpaste was used three times a day to clean the mouth for 12 weeks . Clinical evaluation was using the patient-reported pain score, painkillers, wound healing index (complete epithelization and color matching score), periodontal pocket depth, gingiva index, plaque index and were recorded before operation and 1st, 2nd, 3rd, 4th, 8th, 12th week after surgery. The control group used ordinary toothpaste for oral cleaning, and the rest of the research time, measurement time and measurement results were the same as the experimental group. During the study period, we will continue to monitor whether there is any adverse reaction, and if any adverse reaction occurs, the trial will be stopped.
  Arms: Enoxolone
Other: Sensodyne — The Active Comparator group returned home after the operation and used glycyrrhetinic acid -free toothpaste(Sensodyne) three times a day for oral cleaning. After the operation, toothpaste was used three times a day to clean the mouth for 12 weeks . Clinical evaluation was using the patient-reported pain score, painkillers, wound healing index (complete epithelization and color matching score), periodontal pocket depth, gingiva index, plaque index and were recorded before operation and 1st, 2nd, 3rd, 4th, 8th, 12th week after surgery. The control group used ordinary toothpaste for oral cleaning, and the rest of the research time, measurement time and measurement results were the same as the experimental group. During the study period, we will continue to monitor whether there is any adverse reaction, and if any adverse reaction occurs, the trial will be stopped.
  Arms: Sensodyne

SUMMARY:
Abstract Aim:The Enoxolone (18β-glycyrrhetinic acid; BGA) is a bioactive compound in licorice that exhibits potential anti-ulcer, anti-inflammatory, and anti-microbial activities, relieve oral ulcers, pain, improve gingivitis and dental plaque from past relevant experimental studies,but few clinical trials have evaluated its clinical effectiveness. Therefore, the purpose of this study is to evaluate the effectiveness of Enoxolone on oral conditions of patients with periodontal surgery. Methods:This study is a randomized controlled trial. Patients with severe chronic periodontitis who needed to accept periodontal surgery were randomly assigned to two groups, the experimental group was Enoxolone toothpaste, and the control group for Sensodyne toothpaste. After the operation, toothpaste was used three times a day to clean the mouth for 12 weeks . Clinical evaluation was using the patient-reported pain score, painkillers, wound healing index (complete epithelization and color matching score), periodontal pocket depth, gingiva index, plaque index and were recorded before operation and 1st, 2nd, 3rd, 4th, 8th, 12th week after surgery. Data set performs repeated-measures for the change in mean differences by using the two-tailed independent t tests and generalized linear model.

DETAILED DESCRIPTION:
Enoxolone is a toothpaste containing 18β-glycyrrhetinic acid (BGA). In this study, the experimental group used Enoxolone toothpaste, and the control group did not contain BGA toothpaste (Sensodyne), which is used for oral cleaning of patients after periodontal disease surgery. The absorption rate is very low, and it will not cause any interaction with western medicine.

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 20 years old.
* Those whose health or systemic diseases are well controlled.
* Those with severe chronic periodontitis who need to perform periodontal surgery after being diagnosed by a doctor.
* Subjects who are willing to accept this study.

Exclusion Criteria:

* Allergy to licorice.
* Pregnancy or breastfeeding.
* Periodontal surgery completed at the same site within 6 months.
* Severe bone loss in the apical tissue of the surgical site (including poor prognosis).
* Clinical signs of infection, including fistula, suppuration, fever, severe pain and site swelling.
* Platelets less than 50,000.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
wound healing index | after operation 1st, 2nd, 3rd, 4th, 8th, 12th week
  epithelization and color matching score: A score of 0-10, higher indicates better wound healing.

SECONDARY OUTCOMES:
patient-reported pain score, painkillers | after operation 1week
  the patient-reported pain score(VAS): 0-10 points, the higher the worse. painkillers: 0-15 pills, the more the remaining number of drugs, the better.
Periodontal pocket depth, Gingiva index, Plaque index | after operation 1st, 2nd, 3rd, 4th, 8th, 12th week
  Periodontal pocket depth: 0-15 mm, the higher it means bad. Gingiva index: 0-3 points, higher means bad. Plaque index: 0-3 points, higher means bad.

OTHER OUTCOMES:
adverse event | after operation 1st, 2nd, 3rd, 4th, 8th, 12th week
  allergy

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Tien Hsu, Professor, Study Director — Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No